CLINICAL TRIAL: NCT03580356
Title: A Multi-center, Randomized, Double-blind, Active and Placebo-controlled Study to Investigate the Efficacy and Safety of Ligelizumab (QGE031) in the Treatment of Chronic Spontaneous Urticaria (CSU) in Adolescents and Adults Inadequately Controlled With H1-antihistamines
Brief Title: A Phase III Study of and Efficacy of Ligelizumab in the Treatment of CSU in Adolescents and Adults Inadequately Controlled With H1-antihistamines.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQGE031C2303; 2018-000840-24 (EudraCT Number)
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Results first posted 2024-03-25 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Chronic Spontaneous Urticaria
Keywords: Anti-IgE; CSU; Chronic Spontaneous Urticaria; hives severity score; itch severity score; urticaria activity score
MeSH Terms: conditions — Chronic Urticaria | interventions — ligelizumab; Omalizumab

STUDY DESIGN:
Intervention Model Description: This was a Phase III multi-center, randomized, double-blind, active- and placebo-controlled, parallel-group study. There was a screening period of up to 28 days, a 52 week double-blind treatment period, and a 12 week post-treatment follow-up period.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, investigator staff and personnel performing the study assessments remained blinded to the identity of the treatment from the time of randomization until final database lock. The study drug was prepared by an independent unblinded pharmacist (or authorized delegate) and administered by an independent unblinded study drug administrator. Neither the unblinded pharmacist nor the unblinded study drug administrator was involved in any assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Ligelizumab 120 mg (Experimental): Ligelizumab 120 mg arm: 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
  Interventions: Biological: Ligelizumab
- Ligelizumab 72 mg (Experimental): Ligelizumab 72 mg arm: 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
  Interventions: Biological: Ligelizumab
- Omalizumab 300 mg (Active Comparator): Omalizumab 300 mg arm: 2 injections of 1.2 mL omalizumab q4w
  Interventions: Biological: Omalizumab
- Placebo (Placebo Comparator): Placebo-ligelizumab arm: 2 injections of 1.0mL of ligelizumab placebo from Week 0 through Week 20; 1 injection of 1.0mL of ligelizumab 120 mg + 1 injection of 1.0 mL ligelizumab placebo from Week 24 through Week 48
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Ligelizumab — Liquid in vial
  Arms: Ligelizumab 120 mg; Ligelizumab 72 mg
Biological: Omalizumab — Lyophilized powder for solution in vial
  Arms: Omalizumab 300 mg
Other: Placebo — Liquid in vial
  Arms: Placebo

SUMMARY:
The purpose of this study was to establish efficacy and safety of ligelizumab in adolescent and adult subjects with CSU who remained symptomatic despite standard of care treatment by demonstrating better efficacy over omalizumab and over placebo.

The study population consisted of 1,079 male and female subjects aged ≥ 12 years who were diagnosed with CSU and who remained symptomatic despite the use of H1-antihistamines.

This was a multi-center, randomized, double-blind, active- and placebo-controlled, parallel-group study. There was a screening period of up to 28 days, a 52 week double-blind treatment period, and a 12 week post-treatment follow-up period.

DETAILED DESCRIPTION:
This was a Phase III multi-center, randomized, double-blind, active and placebo-controlled, parallel-group study. The study consisted of 3 distinct periods:

* Screening period (Day -28 to Day 1): Duration of up to 4 weeks in which subjects who have given informed consent were assessed for eligibility.
* Double-blind treatment period (52 weeks): The subjects were seen in the clinic every 4 weeks.
* Post-treatment follow-up period (12 weeks): This period consists of 3 visits (every 4 weeks) with the final visit occurring 16 weeks after the last dose at Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study. The subject's, parent's or legal guardian's signed written informed consent and child's assent, if appropriate, must be obtained before any assessment is performed. Of note, if the subject reaches age of consent (age as per local law) during the study, they will also need to sign the corresponding study Informed Consent Form (ICF) at the next study visit.
* Male and female subjects ≥ 12 years of age at the time of screening.
* CSU diagnosis for ≥ 6 months.
* Diagnosis of CSU refractory to H1-AH at approved doses at the time of randomization, as defined by all of the following:
* The presence of itch and hives for ≥ 6 consecutive weeks at any time prior to Visit 1 (Day - 28 to Day -14) despite current use of non-sedating H1-antihistamine
* UAS7 score (range 0-42) ≥ 16 and HSS7 (range 0-21) ≥ 8 during the 7 days prior to randomization (Visit 110, Day 1)
* Subjects must be on H1-antihistamine at only locally label approved doses for treatment of CSU starting at Visit 1 (Day -28 to Day -14)
* Willing and able to complete a daily symptom eDiary for the duration of the study and adhere to the study visit schedules.

Key Exclusion Criteria:

* History of hypersensitivity to any of the study drugs or their excipients or to drugs of similar chemical classes (i.e. to murine, chimeric or human antibodies).
* Subjects having a clearly defined cause of their chronic urticaria, other than CSU. This includes, but is not limited to, the following: symptomatic dermographism (urticaria factitia), cold-, heat-, solar-, pressure-, delayed pressure-, aquagenic-, cholinergic- or contact-urticaria.
* Diseases, other than chronic urticaria, with urticarial or angioedema symptoms such as urticarial vasculitis, erythema multiforme, cutaneous mastocytosis (urticaria pigmentosa) and hereditary or acquired angioedema (eg, due to C1 inhibitor deficiency).
* Subjects with evidence of helminthic parasitic infection as evidenced by stools being positive for a pathogenic organism according to local guidelines. All subjects will be screened at Visit 1. If stool testing is positive for pathogenic organism, the subject will not be randomized and will not be allowed to rescreen.
* Any other skin disease associated with chronic itching that might influence in the investigators opinion the study evaluations and results (e.g. atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, etc.).
* Prior exposure to ligelizumab or omalizumab.
* H1-AH used as background medication at greater than locally label-approved doses after visit 1

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1078 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (172):
- United States (34):
  - Allervie Clinical Research, Birmingham, Alabama
  - Medical Resch of Arizona-Div of Allergy Asthma and Immunology, Scottsdale, Arizona
  - Atria Clinical Research Asthma and Allergy Institute, Little Rock, Arkansas
  - DeMera Allergy Asthma and Immun Ctr, Fresno, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Jonathan Corren Inc, Los Angeles, California
  - Allergy and Asthma Consultants, Redwood City, California
  - Allergy and Asthma Associates of Santa Clara Vally Center, San Jose, California
  - Sarasota Clinical Research, Sarasota, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Idaho Research, Eagle, Idaho
  - Midwest Allergy Sinus Asthma SC, Normal, Illinois
  - John Hopkins University, Baltimore, Maryland
  - Institute for Asthma and Allergy PC, Chevy Chase, Maryland
  - Chesapeake Clinical Research, White Marsh, Maryland
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Midwest Clinical Research LcLC, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - The Asthma and Allergy Center PC, Papillion, Nebraska
  - Icahn School Of Med At Mount Sinai, New York, New York
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Allergy Asthma and Clinical Research, Oklahoma City, Oklahoma
  - PCR DBA Columbia Asthma and Allergy, Clackamas, Oregon
  - Allergy and Asthma Specialists PC, Blue Bell, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research LLS, North Charleston, South Carolina
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Western Sky Medical Research, El Paso, Texas
  - North Texas Inst For Clinical Tri, Fort Worth, Texas
  - Allergy and Asthma Research Center PA, San Antonio, Texas
  - Quality Assurance Research Center, San Antonio, Texas
  - Allergy and Asthma Care of Waco, Waco, Texas
  - Allergy Associates of Utah, Sandy City, Utah
  - Bellingham Asthma Allergy and Immunology, Bellingham, Washington
- Argentina (7):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Mendoza, Mendoza Province
  - Novartis Investigative Site, Santa Fe, Rosario
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
  - Novartis Investigative Site, Salta
- Australia (3):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, East Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Loverval
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Alphaville Barueri, São Paulo
  - Novartis Investigative Site, São José do Rio Preto, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Chile (3):
  - Novartis Investigative Site, Vitacura, Santiago Metropolitan
  - Novartis Investigative Site, Osorno
  - Novartis Investigative Site, Santiago
- Estonia (2):
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Novartis Investigative Site, Helsinki, Finland
- France (5):
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rouen
- Germany (18):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Halle S
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Quedlinburg
  - Novartis Investigative Site, Simmern
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
- India (5):
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mangalore, Karnataka
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Bikaner, Rajasthan
- Israel (6):
  - Novartis Investigative Site, Afula
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Rehovot
- Italy (6):
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Modena, MO
  - Novartis Investigative Site, Siena, SI
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Chikushino-shi, Fukuoka
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kamimashi-gun, Kumamoto
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Izumo, Shimane
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Machida, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Kobe
- Lebanon (3):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
  - Novartis Investigative Site, Saida
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Villahermosa, Tabasco
- Netherlands (4):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Amersfroort
  - Novartis Investigative Site, Breda
  - Novartis Investigative Site, Utrecht
- Philippines (5):
  - Novartis Investigative Site, Lipa City, Batangas
  - Novartis Investigative Site, City of Taguig, National Capital Region
  - Novartis Investigative Site, Makati City
  - Novartis Investigative Site, Pasig
  - Novartis Investigative Site, Quezon
- Poland (7):
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krosno
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Ossy
  - Novartis Investigative Site, Sopot
  - Novartis Investigative Site, Warsaw
- Romania (5):
  - Novartis Investigative Site, Bucharest, District 2
  - Novartis Investigative Site, Brasov
  - Novartis Investigative Site, Cluj-Napoca
  - Novartis Investigative Site, Craiova
  - Novartis Investigative Site, Iași
- Russia (5):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Stavropol
- Slovakia (8):
  - Novartis Investigative Site, Kežmarok
  - Novartis Investigative Site, Komárno
  - Novartis Investigative Site, Levice
  - Novartis Investigative Site, Nové Zámky
  - Novartis Investigative Site, Považská Bystrica
  - Novartis Investigative Site, Svidník
  - Novartis Investigative Site, Topoľčany
  - Novartis Investigative Site, Žilina
- Spain (10):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Alcorcón, Madrid
  - Novartis Investigative Site, Pozuelo de Alarcón, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Tunisia (3):
  - Novartis Investigative Site, Tunis, Tunisie
  - Novartis Investigative Site, Sfax, Tunusia
  - Novartis Investigative Site, Sousse
- Novartis Investigative Site, London, United Kingdom
- Vietnam (2):
  - Novartis Investigative Site, Hanoi
  - Novartis Investigative Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Maurer M, Ensina LF, Gimenez-Arnau AM, Sussman G, Hide M, Saini S, Grattan C, Fomina D, Rigopoulos D, Berard F, Canonica GW, Rockmann H, Irani C, Szepietowski JC, Leflein J, Bernstein JA, Peter JG, Kulthanan K, Godse K, Ardusso L, Ukhanova O, Staubach P, Sinclair R, Gogate S, Thomsen SF, Tanus T, Ye YM, Burciu A, Barve A, Modi D, Scosyrev E, Hua E, Letzelter K, Varanasi V, Patekar M, Severin T; PEARL-1 and PEARL-2 trial investigators. Efficacy and safety of ligelizumab in adults and adolescents with chronic spontaneous urticaria: results of two phase 3 randomised controlled trials. Lancet. 2024 Jan 13;403(10422):147-159. doi: 10.1016/S0140-6736(23)01684-7. Epub 2023 Nov 23. PMID 38008109

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,078 participants enrolled in 27 countries at 185 sites.
Pre-assignment Details: There were 1,023 adult subjects and 55 adolescent subjects. Out of these 3 adults were mis-randomized and hence did not enter treatment period.
  901 adults and 52 adolescent subjects entered the post treatment follow-up period. The number entering post-treatment follow up is higher than the number completing treatment since this also included subjects who entered the follow up period after early treatment discontinuation.
Groups:
- Ligelizumab 72 mg - Adults; Ligelizumab 72 mg - Adolescents: Ligelizumab 72 mg arm: 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 120 mg - Adults; Ligelizumab 120 mg - Adolescents: Ligelizumab 120 mg arm: 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Omalizumab 300 mg - Adults; Omalizumab 300 mg - Adolescents: Omalizumab 300 mg arm: 2 injections of 1.2 mL omalizumab q4w
- Placebo - Ligelizumab 120mg - Adults; Placebo - Ligelizumab 120mg - Adolescents: 2 injections of 1.0 mL of ligelizumab placebo q4w from Week 0 to Week 20; 1.0 mL of ligelizumab 120 mg + 1.0 mL of ligelizumab placebo q4w from Week 24 through Week 48
Period: Treatment Period
Arm/Group | Ligelizumab 72 mg - Adults | Ligelizumab 72 mg - Adolescents | Ligelizumab 120 mg - Adults | Ligelizumab 120 mg - Adolescents | Omalizumab 300 mg - Adults | Omalizumab 300 mg - Adolescents | Placebo - Ligelizumab 120mg - Adults | Placebo - Ligelizumab 120mg - Adolescents
Started | 307 | 16 | 304 | 19 | 309 | 14 | 103 | 6
Randomized Set (RAN) | 307 | 16 | 304 | 19 | 309 | 14 | 103 | 6
Safety Set (SAF) | 304 | 16 | 306 | 19 | 307 | 14 | 103 | 6
Full Analysis Set (FAS) | 307 | 16 | 303 | 19 | 307 | 14 | 103 | 6
Completed | 269 | 15 | 259 | 17 | 263 | 13 | 82 | 6
Not Completed | 38 | 1 | 45 | 2 | 46 | 1 | 21 | 0
Not completed — Withdrawal by Subject | 13 | 0 | 13 | 1 | 17 | 0 | 5 | 0
Not completed — Adverse Event | 10 | 0 | 13 | 0 | 5 | 0 | 8 | 0
Not completed — Protocol Violation | 5 | 0 | 6 | 1 | 9 | 1 | 1 | 0
Not completed — Lack of Efficacy | 6 | 0 | 2 | 0 | 3 | 0 | 3 | 0
Not completed — Pregnancy | 1 | 0 | 7 | 0 | 2 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 1 | 0 | 4 | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Technical problems | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Misrandomized, no treatment | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Period: Post-treatment Follow Up Period
Arm/Group | Ligelizumab 72 mg - Adults | Ligelizumab 72 mg - Adolescents | Ligelizumab 120 mg - Adults | Ligelizumab 120 mg - Adolescents | Omalizumab 300 mg - Adults | Omalizumab 300 mg - Adolescents | Placebo - Ligelizumab 120mg - Adults | Placebo - Ligelizumab 120mg - Adolescents
Started (Entered post-treatment follow up period) | 272 | 15 | 275 | 18 | 265 | 13 | 89 | 6
Completed | 260 | 15 | 256 | 17 | 259 | 13 | 82 | 5
Not Completed | 12 | 0 | 19 | 1 | 6 | 0 | 7 | 1
Not completed — Withdrawal by Subject | 6 | 0 | 12 | 1 | 4 | 0 | 6 | 1
Not completed — Lost to Follow-up | 3 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to.
Groups:
- Placebo: Placebo-ligelizumab arm: 2 injections of 1.0mL of ligelizumab placebo from Week 0 through Week 20
- Total: Total of all reporting groups
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo | Total
Number analyzed (Participants) | 323 | 323 | 323 | 109 | 1078
Age, Categorical [Count of Participants; unit: Participants] — Population: Randomized Set
  Participants
    Adults: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adults: <=18 years | 0 | 0 | 0 | 0 | 0
    Adults: Between 18 and 65 years | 288 | 278 | 286 | 96 | 948
    Adults: >=65 years | 19 | 26 | 23 | 7 | 75
    Adolescents: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescents: <=18 years | 16 | 19 | 14 | 6 | 55
    Adolescents: Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
    Adolescents: >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to.
  Years
    Adults: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adults | 41.7 (13.42) | 43.0 (14.11) | 44.1 (14.11) | 42.9 (13.01) | 42.9 (13.81)
    Adolescents: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescents | 14.3 (1.39) | 15.1 (1.56) | 15.9 (1.17) | 14.8 (1.47) | 15.0 (1.50)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to.
  Participants
    Adult: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult: Female | 227 | 211 | 225 | 80 | 743
    Adult: Male | 80 | 93 | 84 | 23 | 280
    Adolescent: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent: Female | 10 | 12 | 10 | 4 | 36
    Adolescent: Male | 6 | 7 | 4 | 2 | 19
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Randomized set (RAN) included all randomized subjects, regardless of whether or not they received a dose of study drug. Subjects were analyzed according to the treatment they were assigned to.
  Participants
    Adult White: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult White | 227 | 218 | 228 | 79 | 752
    Adolescent White: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent White | 9 | 15 | 10 | 5 | 39
    Adult Black or African American: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult Black or African American | 5 | 12 | 9 | 1 | 27
    Adolescent Black or African American: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent Black or African American | 1 | 0 | 0 | 0 | 1
    Adult Asian: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult Asian | 66 | 67 | 63 | 19 | 215
    Adolescent Asian: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent Asian | 2 | 2 | 4 | 0 | 8
    Adult Native Hawaiian or Other Pacific Islander: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Adolescent Native Hawaiian or Pacific Islander: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
    Adult Native American: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult Native American | 7 | 4 | 6 | 3 | 20
    Adolescents Native American: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescents Native American | 4 | 2 | 0 | 1 | 7
    Adult Multi-racial: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult Multi-racial | 2 | 3 | 3 | 1 | 9
    Adolescent Multi-racial: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent Multi-racial | 0 | 0 | 0 | 0 | 0
    Adult Race Not Reported: number analyzed (Participants) | 307 | 304 | 309 | 103 | 1023
    Adult Race Not Reported | 0 | 0 | 0 | 0 | 0
    Adolescent Race Not Reported: number analyzed (Participants) | 16 | 19 | 14 | 6 | 55
    Adolescent Race Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Number and Percentage of Subjects With UAS7=0 Response at Week 12 (Multiple Imputation - Adults, Observed Data for Adolescents)
Description: The Urticaria Activity Score (UAS) is the sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is the sum of the HSS7 and the ISS7 scores. The possible range of the weekly UAS7 score is 0 to 42. Complete UAS7 response is defined as UAS7 = 0. Data is presented as percentage of patients with a UAS7=0 score. No Statistical analysis was planned for adolescent group.
Time Frame: Week 12
Population: FAS: Adults + Adolescents = Total
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 322 | 320 | 321 | 109
Participants
  Adults: number analyzed (Participants) | 307 | 303 | 307 | 103
  Adults | 88 | 103 | 94 | 4
  Adolescents: number analyzed (Participants) | 15 | 17 | 14 | 6
  Adolescents | 4 | 8 | 5 | 0
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 9.029, 95% CI 2-sided [3.183 to 25.615]
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.6646, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 0.926, 95% CI 2-sided [0.650 to 1.319]
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 11.508, 95% CI 2-sided [4.058 to 32.638]
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.1730, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio, log = 1.181, 95% CI 2-sided [0.836 to 1.667]

2. Primary Outcome: Mean Change From Baseline in UAS7 at Week 12 (Multiple Imputation) of Adult Subjects
Description: The Urticaria Activity Score (UAS) is sum of the Hive Severity Score (HSS) and the Itch Severity Score (ISS). UAS7 is sum of the HSS7 and the ISS7 scores. Possible range of weekly UAS7 score is 0 to 42. Complete UAS7 response is UAS7 = 0. Hives Severity Score (HSS) scale is 0 to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. Possible range of the weekly score is therefore 0 to 21. Hives Severity Score scale: 0 - None 1 - Mild (1-6 hives/12 hours) 2 - Moderate (7-12 hives/12 hours) 3 - Severe (>12 hives/12 hours). Itch Severity Score (ISS) scale is 0 to 3. Score (ISS7) is derived by adding up average daily scores of 7 days preceding visit. Possible range of weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate). Negative change from baseline indicates improvement
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized Adult subjects who received at least one dose of study drug. Subjects were analyzed according to the treatment to which they were assigned at randomization. FAS was used for all efficacy variables, unless otherwise stated.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 307 | 303 | 307 | 103
Scores on a scale | -19.218 (0.651) | -20.312 (0.654) | -19.632 (0.652) | -9.221 (1.135)
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Treatment contrast in LS mean (change), Adults only; Test type: Superiority; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -9.997, 95% CI 2-sided [-12.554 to -7.439], Standard Error of Mean 1.305
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Treatment contrast in LS mean (change), Adults only; Test type: Superiority; p = 0.6735, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS mean = 0.414, 95% CI 2-sided [-1.392 to 2.221], Standard Error of Mean 0.922
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Treatment contrast in LS mean (change), Adults only; Test type: Superiority; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -11.091, 95% CI 2-sided [-13.664 to -8.518], Standard Error of Mean 1.313
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Treatment contrast in LS mean (change), Adults only; Test type: Superiority; p = 0.2305, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS mean = -0.680, 95% CI 2-sided [-2.489 to 1.128], Standard Error of Mean 0.923

3. Primary Outcome: Mean Change From Baseline in UAS7 at Week 12 (Observed Data) of Adolescent Subjects (FAS)
Description: as for outcome 2
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS) included all randomized adolescent subjects who received at least one dose of study drug. Subjects were analyzed according to the treatment to which they were assigned at randomization. FAS was used for all efficacy variables, unless otherwise stated.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 16 | 19 | 14 | 6
scores on a scale | -14.92 (13.479) | -24.83 (12.640) | -18.16 (10.246) | -11.94 (14.278)

4. Secondary Outcome: Mean Change From Baseline in ISS7 at Week 12 (Multiple Imputation) of Adult Subjects (FAS)
Description: Improvement of severity of itch assessed as absolute change from baseline in ISS7 score at Week 12 Itch Severity Score (ISS) is on a scale of 0 to 3. A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate) Negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12
Population: FAS: Adults
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 307 | 303 | 307 | 103
scores on a scale | -8.632 (0.298) | -9.023 (0.300) | -8.733 (0.300) | -4.527 (0.522)
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults only; Test type: Superiority; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -4.105, 95% CI 2-sided [-5.281 to -2.929], Standard Error of Mean 0.600
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority; p = 0.5943, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = 0.101, 95% CI 2-sided [-0.727 to 0.928], Standard Error of Mean 0.422
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Test type: Superiority — Adults only; p < .0001, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -4.496, 95% CI 2-sided [-5.678 to -3.314], Standard Error of Mean 0.603
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority; p = 0.2467, Mixed Models Analysis; Linear mixed model with repeated measures (MMRM); LS Mean = -0.290, 95% CI 2-sided [-1.120 to 0.540], Standard Error of Mean 0.423

5. Secondary Outcome: Mean Change From Baseline in ISS7 at Week 12 (Observed Data) of Adolescent Subjects, (FAS)
Description: Improvement of severity of itch assessed as absolute change from baseline in ISS7 score at Week 12 Itch Severity Score (ISS) is on a scale of 0 to 3. A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 to 21. Itch Severity Score scale: 0 - None 1 - Mild (minimal awareness, easily tolerated) 2 - Moderate (definite awareness, bothersome but tolerable) 3 - Severe (difficult to tolerate) Negative change from baseline indicates improvement.. No Statistical Analysis was planned for adolescent population.
Time Frame: Baseline, Week 12
Population: FAS: Adolescents
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 16 | 19 | 14 | 6
scores on a scale | -6.38 (6.994) | -12.04 (6.264) | -8.56 (4.935) | -6.97 (7.904)

6. Secondary Outcome: Number and Percentage of Participants With DLQI Score of 0 - 1 at Week 12 (Multiple Imputation - Adults, Observed Data for Adolescents)
Description: Assessed as percentage of subjects achieving DLQI = 0-1, which means No impact on subjects quality of life at Week 12 The Dermatology life Quality Index (DLQI) score range is 0 to 30, with 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life). Data is presented as percentage of patients with a DLQI=0 score. No statistical analysis was planned for adolescent group.
Time Frame: Week 12
Population: FAS: Adults + Adolescents = Total
Measure: Count of Participants; unit: Participants
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 322 | 319 | 319 | 109
Participants
  Adults: number analyzed (Participants) | 307 | 303 | 307 | 103
  Adults | 134 | 153 | 147 | 18
  Adolescents: number analyzed (Participants) | 15 | 16 | 12 | 6
  Adolescents | 4 | 9 | 5 | 0
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 3.443, 95% CI 2-sided [1.955 to 6.063]
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.8524, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 0.838, 95% CI 2-sided [0.602 to 1.167]
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p < .0001, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 4.542, 95% CI 2-sided [2.577 to 8.004]
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority — Wald chi-square test based on logistic regression; p = 0.2764, Regression, Logistic; 95% confidence interval for the odds ratio; Odds Ratio (OR) = 1.106, 95% CI 2-sided [0.794 to 1.540]

7. Secondary Outcome: Cumulative Number of Weeks of AAS7=0 up to Week 12 (Multiple Imputation) of Adult Subjects (FAS)
Description: Cumulative number of weeks that subjects achieve AAS7 = 0 responses between baseline and Week 12 Angioedema Activity Score (AAS7) is a measure of the frequency and intensity of angioedema episodes. The total possible range of scores over 7 days is 0-15 (mean day sum score) where higher scores indicate increased angioedema activity.
Time Frame: Baseline, Week 12
Population: FAS: Adults
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 307 | 303 | 307 | 103
Weeks | 8.668 (0.241) | 8.897 (0.246) | 8.427 (0.237) | 6.242 (0.331)
Statistical Analysis 1: Comparison: Ligelizumab 72 mg vs Placebo; Adults only; Test type: Superiority; p < .0001, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.389, 95% CI 2-sided [1.235 to 1.561]
Statistical Analysis 2: Comparison: Ligelizumab 72 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority; p = 0.2369, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.029, 95% CI 2-sided [0.952 to 1.111]
Statistical Analysis 3: Comparison: Ligelizumab 120 mg vs Placebo; Adults only; Test type: Superiority; p < .0001, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.425, 95% CI 2-sided [1.268 to 1.603]
Statistical Analysis 4: Comparison: Ligelizumab 120 mg vs Omalizumab 300 mg; Adults only; Test type: Superiority; p = 0.0830, Negative binomial regression model; 95% confidence interval for the relative risk ratio; Risk Ratio (RR) = 1.056, 95% CI 2-sided [0.978 to 1.140]

8. Secondary Outcome: Cumulative Number of Weeks of AAS7=0 up to Week 12 (Observed Data) of Adolescent Subjects (FAS)
Description: Cumulative number of weeks that subjects achieve AAS7 = 0 responses between baseline and Week 12 Angioedema Activity Score (AAS7) is a measure of the frequency and intensity of angioedema episodes. The total possible range of scores over 7 days is 0-15 (mean day sum score) where higher scores indicate increased angioedema activity. No Statistical Analysis was planned.
Time Frame: Baseline, Week 12
Population: FAS: Adolescents
Measure: Least Squares Mean (Standard Error); unit: Weeks
Arm/Group | Ligelizumab 72 mg | Ligelizumab 120 mg | Omalizumab 300 mg | Placebo
Number analyzed (Participants) | 16 | 19 | 14 | 6
Weeks | 6.8 (4.90) | 8.6 (4.60) | 10.2 (3.01) | 9.2 (4.92)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) monitoring was continued for at least 30 days following the last dose of study treatment or end of study visit (64 weeks), whichever was longer.
Groups:
- Ligelizumab 72mg (Adults): Ligelizumab 72mg (Adults): 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 72mg (Adolescents): Ligelizumab 72mg (Adolescents): 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 72mg (Adults+Adolescents): Ligelizumab 72mg (Adults+Adolescents): 1 injection of 0.6 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 120 mg (Adults): Ligelizumab 120 mg (Adults): 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 120 mg (Adolescents): Ligelizumab 120 mg (Adolescents): 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Ligelizumab 120 mg (Adults+Adolescents): Ligelizumab 120 mg (Adults+Adolescents): 1 injection of 1.0 mL ligelizumab + 1 injection of 1.0 mL ligelizumab placebo q4w
- Omalizumab 300mg (Adults): Omalizumab 300mg (Adults): 2 injections of 1.2 mL omalizumab q4w
- Omalizumab 300mg (Adolescents): Omalizumab 300mg (Adolescents): 2 injections of 1.2 mL omalizumab q4w
- Omalizumab 300mg (Adults+Adolescents): Omalizumab 300mg (Adults+Adolescents): 2 injections of 1.2 mL omalizumab q4w
- Placebo Only (Adults): Placebo only (Adults): Safety events between Wk 0- 24 (until participants received Ligelizumab 120 mg) are presented
- Placebo Only (Adolescents): Placebo only (Adolescents): Safety events between Wk 0- 24 (until participants received Ligelizumab 120 mg) are presented
- Placebo Only (Adults+Adolescents): Placebo only (Adults+Adolescents): Safety events between Wk 0- 24 (until participants received Ligelizumab 120 mg) are presented
- Transitioned to Ligelizumab 120mg (Adults): Placebo Adults patients who transitioned to ligelizumab 120mg; 1 injection of 1.0mL of ligelizumab, 120 mg + 1 injection of 1.0 mL ligelizumab placebo from Week 24 through Week 48. At week 24 participants received active drug. Safety events from week 24 to end of study are presented.
- Transitioned to Ligelizumab 120mg (Adolescents): Placebo Adolescents patients who transitioned to ligelizumab 120mg; 1 injection of 1.0mL of ligelizumab, 120 mg + 1 injection of 1.0 mL ligelizumab placebo from Week 24 through Week 48. At week 24 participants received active drug. Safety events from week 24 to end of study are presented.
- Transitioned to Ligelizumab 120mg (Adults+Adolescents): Placebo Adults+Adolescents patients who transitioned to ligelizumab 120mg; 1 injection of 1.0mL of ligelizumab, 120 mg + 1 injection of 1.0 mL ligelizumab placebo from Week 24 through Week 48. At week 24 participants received active drug. Safety events from week 24 to end of study are presented.
Arm/Group | Ligelizumab 72mg (Adults) | Ligelizumab 72mg (Adolescents) | Ligelizumab 72mg (Adults+Adolescents) | Ligelizumab 120 mg (Adults) | Ligelizumab 120 mg (Adolescents) | Ligelizumab 120 mg (Adults+Adolescents) | Omalizumab 300mg (Adults) | Omalizumab 300mg (Adolescents) | Omalizumab 300mg (Adults+Adolescents) | Placebo Only (Adults) | Placebo Only (Adolescents) | Placebo Only (Adults+Adolescents) | Transitioned to Ligelizumab 120mg (Adults) | Transitioned to Ligelizumab 120mg (Adolescents) | Transitioned to Ligelizumab 120mg (Adults+Adolescents)
All-Cause Mortality (participants affected / at risk) | 0/304 | 0/16 | 0/320 | 1/306 | 0/19 | 1/325 | 0/307 | 0/14 | 0/321 | 0/103 | 0/6 | 0/109 | 0/90 | 0/6 | 0/96
Serious Adverse Events (participants affected / at risk) | 3/304 | 0/16 | 3/320 | 3/306 | 0/19 | 3/325 | 2/307 | 0/14 | 2/321 | 1/103 | 0/6 | 1/109 | 0/90 | 0/6 | 0/96
Other Adverse Events (participants affected / at risk) | 177/304 | 7/16 | 184/320 | 182/306 | 10/19 | 192/325 | 165/307 | 10/14 | 175/321 | 40/103 | 1/6 | 41/109 | 37/90 | 2/6 | 39/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 72mg (Adults) (N=304) | Ligelizumab 72mg (Adolescents) (N=16) | Ligelizumab 72mg (Adults+Adolescents) (N=320) | Ligelizumab 120 mg (Adults) (N=306) | Ligelizumab 120 mg (Adolescents) (N=19) | Ligelizumab 120 mg (Adults+Adolescents) (N=325) | Omalizumab 300mg (Adults) (N=307) | Omalizumab 300mg (Adolescents) (N=14) | Omalizumab 300mg (Adults+Adolescents) (N=321) | Placebo Only (Adults) (N=103) | Placebo Only (Adolescents) (N=6) | Placebo Only (Adults+Adolescents) (N=109) | Transitioned to Ligelizumab 120mg (Adults) (N=90) | Transitioned to Ligelizumab 120mg (Adolescents) (N=6) | Transitioned to Ligelizumab 120mg (Adults+Adolescents) (N=96)
COVID-19 (Infections and infestations) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ligelizumab 72mg (Adults) (N=304) | Ligelizumab 72mg (Adolescents) (N=16) | Ligelizumab 72mg (Adults+Adolescents) (N=320) | Ligelizumab 120 mg (Adults) (N=306) | Ligelizumab 120 mg (Adolescents) (N=19) | Ligelizumab 120 mg (Adults+Adolescents) (N=325) | Omalizumab 300mg (Adults) (N=307) | Omalizumab 300mg (Adolescents) (N=14) | Omalizumab 300mg (Adults+Adolescents) (N=321) | Placebo Only (Adults) (N=103) | Placebo Only (Adolescents) (N=6) | Placebo Only (Adults+Adolescents) (N=109) | Transitioned to Ligelizumab 120mg (Adults) (N=90) | Transitioned to Ligelizumab 120mg (Adolescents) (N=6) | Transitioned to Ligelizumab 120mg (Adults+Adolescents) (N=96)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 5 | 0 | 5 | 8 | 0 | 8 | 1 | 0 | 1 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 0 | 11 | 10 | 0 | 10 | 6 | 1 | 7 | 4 | 0 | 4 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 9 | 2 | 11 | 4 | 0 | 4 | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 11 | 1 | 12 | 11 | 0 | 11 | 8 | 0 | 8 | 1 | 0 | 1 | 3 | 0 | 3
Gastritis (Gastrointestinal disorders) | 4 | 0 | 4 | 3 | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 0 | 7 | 2 | 0 | 2 | 3 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 13 | 2 | 15 | 10 | 1 | 11 | 8 | 1 | 9 | 2 | 0 | 2 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 4 | 0 | 4 | 5 | 0 | 5 | 8 | 0 | 8 | 4 | 0 | 4 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 10 | 1 | 11 | 7 | 0 | 7 | 4 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 8 | 2 | 10 | 9 | 0 | 9 | 7 | 0 | 7 | 1 | 0 | 1 | 1 | 0 | 1
Injection site erythema (General disorders) | 7 | 1 | 8 | 12 | 0 | 12 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 2
Injection site pain (General disorders) | 6 | 1 | 7 | 5 | 1 | 6 | 5 | 0 | 5 | 1 | 0 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 5 | 0 | 5 | 8 | 1 | 9 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1
Injection site swelling (General disorders) | 6 | 0 | 6 | 5 | 1 | 6 | 1 | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 3
Injection site urticaria (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Pyrexia (General disorders) | 6 | 2 | 8 | 8 | 1 | 9 | 10 | 0 | 10 | 0 | 0 | 0 | 2 | 0 | 2
Bronchitis (Infections and infestations) | 8 | 0 | 8 | 3 | 1 | 4 | 9 | 0 | 9 | 1 | 0 | 1 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 17 | 0 | 17 | 16 | 2 | 18 | 10 | 2 | 12 | 1 | 0 | 1 | 4 | 0 | 4
Gastroenteritis (Infections and infestations) | 9 | 0 | 9 | 6 | 0 | 6 | 7 | 0 | 7 | 1 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 14 | 2 | 16 | 11 | 2 | 13 | 9 | 0 | 9 | 1 | 0 | 1 | 3 | 0 | 3
Nasopharyngitis (Infections and infestations) | 42 | 2 | 44 | 36 | 3 | 39 | 36 | 4 | 40 | 6 | 1 | 7 | 7 | 0 | 7
Oral herpes (Infections and infestations) | 1 | 0 | 1 | 5 | 0 | 5 | 4 | 0 | 4 | 3 | 0 | 3 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 4 | 0 | 4 | 4 | 0 | 4 | 3 | 0 | 3 | 1 | 0 | 1 | 1 | 1 | 2
Sinusitis (Infections and infestations) | 2 | 1 | 3 | 5 | 0 | 5 | 7 | 1 | 8 | 2 | 0 | 2 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 2 | 4 | 0 | 4 | 7 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 17 | 0 | 17 | 17 | 2 | 19 | 15 | 0 | 15 | 1 | 0 | 1 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 0 | 4 | 11 | 0 | 11 | 18 | 0 | 18 | 0 | 0 | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 1 | 4 | 3 | 0 | 3 | 10 | 0 | 10 | 2 | 0 | 2 | 0 | 0 | 0
SARS-CoV-2 test negative (Investigations) | 7 | 0 | 7 | 1 | 1 | 2 | 4 | 0 | 4 | 1 | 0 | 1 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 0 | 8 | 15 | 0 | 15 | 14 | 0 | 14 | 1 | 0 | 1 | 3 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 0 | 19 | 20 | 1 | 21 | 15 | 0 | 15 | 2 | 0 | 2 | 2 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 1 | 6 | 8 | 1 | 9 | 1 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 1 | 7 | 3 | 0 | 3 | 7 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 35 | 4 | 39 | 44 | 2 | 46 | 37 | 2 | 39 | 7 | 0 | 7 | 6 | 0 | 6
Migraine (Nervous system disorders) | 1 | 0 | 1 | 4 | 0 | 4 | 3 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 3
Somnolence (Nervous system disorders) | 3 | 0 | 3 | 4 | 0 | 4 | 1 | 2 | 3 | 3 | 0 | 3 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 8 | 1 | 9 | 4 | 0 | 4 | 2 | 0 | 2 | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 7 | 12 | 0 | 12 | 5 | 1 | 6 | 2 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 13 | 9 | 1 | 10 | 4 | 1 | 5 | 2 | 0 | 2 | 2 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 0 | 3 | 9 | 1 | 10 | 5 | 1 | 6 | 0 | 0 | 0 | 1 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 13 | 1 | 14 | 6 | 0 | 6 | 8 | 0 | 8 | 1 | 0 | 1 | 1 | 0 | 1
Chronic spontaneous urticaria (Skin and subcutaneous tissue disorders) | 8 | 1 | 9 | 8 | 0 | 8 | 4 | 0 | 4 | 1 | 0 | 1 | 2 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 | 0 | 5 | 9 | 0 | 9 | 3 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 12 | 0 | 12 | 12 | 0 | 12 | 10 | 2 | 12 | 1 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 13 | 0 | 13 | 17 | 0 | 17 | 11 | 1 | 12 | 4 | 0 | 4 | 1 | 1 | 2
Hypertension (Vascular disorders) | 11 | 0 | 11 | 10 | 0 | 10 | 9 | 0 | 9 | 0 | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-01-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT03580356/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03580356/SAP_001.pdf